CLINICAL TRIAL: NCT06450886
Title: An Open-label, Multicenter Study to Evaluate the Long-term Safety and Efficacy of Ulviprubart (ABC008) in Subjects Who Have Completed a Trial of Ulviprubart for the Treatment of Inclusion Body Myositis
Brief Title: Long-term Extension Study of Ulviprubart (ABC008) in Subjects With Inclusion Body Myositis
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Abcuro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABC008-IBM-202
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2024-10

CONDITIONS: Inclusion Body Myositis (IBM)
MeSH Terms: conditions — Myositis, Inclusion Body

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ulviprubart (ABC008) 2.0 mg/kg SC (Experimental): All eligible subjects, regardless of treatment assignment or dose level in their initial study, will be administered ulviprubart at a dose of 2.0 mg/kg via subcutaneous (SC) injection Q8W.
  Interventions: Drug: Ulviprubart (ABC008)

INTERVENTIONS:
Drug: Ulviprubart (ABC008) — All eligible subjects, regardless of treatment assignment or dose level in their initial study, will be administered ulviprubart at a dose of 2.0 mg/kg via subcutaneous (SC) injection Q8W.

SUMMARY:
ABC008-IBM-202 is an open-label, multicenter study to evaluate the safety and efficacy of long-term administration of ulviprubart (ABC008) in subjects with IBM who have completed either Study ABC008-IBM-101 or Study ABC008-IBM-201. Subjects may be enrolled in this study if they meet study eligibility criteria and:

* Have completed the Part 2 (Multiple Ascending Dose [MAD]) End of-Treatment (EOT) Visit in Study ABC008-IBM-101; subjects who continued further on into Part 3 of the study (MAD Extension) prior to enrolling in this study are also eligible; OR
* Have completed the Week 80 Follow-up Visit in Study ABC008-IBM-201.

DETAILED DESCRIPTION:
ABC008-IBM-202 is an open-label, multicenter study to evaluate the safety and efficacy of long-term administration of ulviprubart (ABC008) in subjects with IBM who have completed either Study ABC008-IBM-101 or Study ABC008-IBM-201. Subjects may be enrolled in this study if they meet study eligibility criteria and:

* Have completed the Part 2 (Multiple Ascending Dose [MAD]) End of-Treatment (EOT) Visit in Study ABC008-IBM-101; subjects who continued further on into Part 3 of the study (MAD Extension) prior to enrolling in this study are also eligible; OR
* Have completed the Week 80 Follow-up Visit in Study ABC008-IBM-201. Subjects will enter this study following their initial study such that dosing continues every eight weeks (Q8W) between the last dose in the initial study and the first dose in this long-term extension (LTE) Study IBM-202. Study subjects will continue to receive any ongoing concomitant medications from the initial study.

Subjects will be required to sign an informed consent form before undertaking any study-specific procedures or assessments. Screening is intended to be done at the final visit of the initial study, which will coincide with the Baseline (Day 1) Visit for this study; if this is not possible, the Baseline (Day 1) Visit for this study, including screening, may be conducted at a separate visit (provided it occurs within the visit window defined in Appendix 1 of the protocol). Subsequent study visits will occur every eight weeks until EOT at Week 156, or withdrawal from the study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Able to read, understand, and provide signed informed consent prior to the performance of any study-related procedures.

  2. Has participated in and completed either Study ABC008-IBM-101 or Study ABC008-IBM-201; completion of the prior study will be defined as completion of the Part 2 (MAD) EOT Visit in Study ABC008-IBM-101 (subjects may have continued into Part 3 [MAD Extension]) or completion of the Week 80 Follow-up Visit in Study ABC008-IBM-201.

  3. Demonstrated adequate compliance, in the opinion of the Investigator, with the study procedures during Study ABC008-IBM-101 or Study ABC008-IBM-201.

  4. Willing and able to comply with the requirements of the protocol, including traveling to the site for study-related assessments and SC injections of ulviprubart.

  5. Women of childbearing potential (WOCBP) and male subjects with female partners who are WOCBP (based on sex assignation at birth) must agree to use highly effective (< 1% failure rate) contraception for the duration of the study through 180 days after EOT/ETV.

  6. WOCBP (based on sex assignation at birth) must have a negative urine pregnancy test at the Baseline (Day 1) Visit.

  7. Male subjects (based on sex assignation at birth) must refrain from sperm donation for the duration of the study through 180 days after EOT/ETV.

Exclusion Criteria:

* 1. Has an unresolved clinically significant AE or a clinically significant finding on a clinical laboratory test, ECG, or physical examination during Study ABC008-IBM-101 or Study ABC008 IBM-201 that, in the Investigator's opinion, would limit the subject's ability to participate in or comply with this study.

  2. Participation in another investigational drug study (other than Study ABC008-IBM-101 or Study ABC008-IBM-201) within 30 days prior to the Baseline (Day 1) Visit or five times the half-life of the investigational drug, whichever is longer.

  3. Is not willing or able to comply with the restrictions regarding the use of prohibited medications throughout the study.

  4. Women who are pregnant, lactating, or who plan to become pregnant or initiate lactation during the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | From Baseline (Day 1) through study completion, an average of 156 weeks.]
  The primary endpoint for the study will be the incidence, type, and severity of treatment-emergent adverse events (TEAEs). Safety as assessed by the incidence, type and severity of Treatment Emergent Adverse Events (TEAEs)

SECONDARY OUTCOMES:
Treatment Emergent Serious Adverse Events (TEASAEs) | From Baseline (Day 1) through study completion, an average of 156 weeks.]
  Incidence, type, and severity of treatment-emergent serious adverse events (TESAEs)
Treatment Emergent Adverse Events (TEAEs) onset within 24 hours of Study Medication Administration. | From Baseline (Day 1) through study completion, an average of 156 weeks.]
  Incidence of TEAEs leading to study medication or study discontinuation
Adverse Events of Special Interest (AESI) | From Baseline (Day 1) through study completion, an average of 156 weeks.]
  Incidence of Adverse events of special interest (AESIs)
Change from baseline standard laboratory parameters (Hematology) | From Baseline (Day 1) through study completion, an average of 156 weeks.]
  Incidence of clinically significant changes in standard laboratory parameters (Hematology)
Change from baseline in standard laboratory parameters (Chemistry) | From Baseline (Day 1) through study completion, an average of 156 weeks.]
  Incidence of clinically significant changes from baseline in standard laboratory parameters (Chemistry)
Change from baseline in standard laboratory parameters (Coagulation) | From Baseline (Day 1) through study completion, an average of 156 weeks.]
  Incidence of clinically significant changes from baseline standard laboratory parameters (Coagulation)
Inclusion Body Myositis Functional Rating Scale (IBMFRS) | From Baseline (Day 1) through study completion, an average of 156 weeks.]
  Mean change from Baseline (Day 1) in IBMFRS over the duration of the study
Manual Muscle Test 12 (MMT 12) | From Baseline (Day 1) through study completion, an average of 156 weeks.]
  Mean change from Baseline (Day 1) in MMT 12 over the duration of the study
Change from baseline in standard vital signs (respiratory rate) | From Baseline (Day 1) through study completion, an average of 156 weeks.]
  Incidence of clinically significant changes in vital signs (respiratory rate)
Change from baseline in standard vital signs blood pressure | From Baseline (Day 1) through study completion, an average of 156 weeks.]
  Incidence of clinically significant changes in standard vital signs blood pressure (Systolic and diastolic) blood pressure)
Change from baseline in standard vital signs (temperature) | From Baseline (Day 1) through study completion, an average of 156 weeks.]
  Incidence of clinically significant changes in standard vital signs (temperature)
Change from baseline in standard vital signs (pulse rate) | From Baseline (Day 1) through study completion, an average of 156 weeks.]
  Incidence of clinically significant changes in standard vital signs (pulse rate)
Counts of absolute and KLRG1+ lymphocytes by flow cytometry. | From Baseline (Day 1) through study completion, an average of 156 weeks.]
  Blood samples will be collected for immunophenotyping. Counts of absolute and KLRG1+ lymphocytes and other lymphocyte subsets will be performed by flow cytometry.
Presence and titer of antidrug antibodies (ADA) | From Baseline (Day 1) through study completion, an average of 156 weeks.]
  The incidence and titers of ADAs to ulviprubart will be evaluated in blood samples
Serum concentration of ulviprubart | From Baseline (Day 1) through study completion, an average of 156 weeks.]
  Individual and mean serum concentration time profiles will be presented graphically using nominal time points.

CONTACTS AND LOCATIONS:
Locations (21):
- United States (18):
  - Neuromuscular Research Center, Phoenix, Arizona
  - University of California Irvine Medical Center (UCIMC) - Amyotrophic Lateral Sclerosis (ALS) and Neuromuscular Center, Irvine, California
  - Keck Hospital of USC, Los Angeles, California
  - Yale School of Medicine, New Haven, Connecticut
  - Neuromuscular Diagnostic Center - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Hospital for Special Surgery, New York, New York
  - Duke Neurological Disorders Clinic, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Arthritis and Autoimmunity Center, Falk Clinic, Pittsburgh, Pennsylvania
  - Austin Neuromuscular Center, Austin, Texas
  - Texas Neurology, Dallas, Texas
  - Nerve and Muscle Center of Texas, Houston, Texas
  - Virginia Commonwealth University, Henrico, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Perron Institute for Neurological and Translational Science, Nedlands, Washington

IPD SHARING:
Plan to Share IPD: Undecided